CLINICAL TRIAL: NCT02459067
Title: Adaptive Study of the Safety, Tolerability & Efficacy of Autologous γδ T Lymphocyte Therapy (ImmuniCell®) in Patients With Advanced Cancers Refractory to Current Treatment or Have Indolent Disease for Which Immunotherapy May be Beneficial
Brief Title: ImmuniCell® in Patients With Advanced Cancers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: TC Biopharm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCB-101-001
Record Dates: First submitted 2015-05-20; First posted 2015-06-01 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Malignant Melanoma; Non-small Cell Lung Cancer; Renal Cell Cancer
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ImmuniCell® (Experimental): Subjects will receive 6 cycles of ImmuniCell®, one infusion over an hour, at two-week intervals. During Stage 1, intra-patient dose escalation to achieve a total dose of 30 x 109 γδ T cells.
  Interventions: Biological: ImmuniCell®

INTERVENTIONS:
Biological: ImmuniCell® — Autologous γδ T Lymphocytes

SUMMARY:
To determine the safety, tolerability, maximum tolerated dose (MTD) and efficacy of ImmuniCell® in patients with melanoma, renal cell cancer (RCC) or non-small cell lung cancer (NSCLC). The study is an adaptive design that has 3 stages: Stage 1 - dose escalation, Stage 2 - efficacy, and Stage 3 - confirm efficacy in one of the tumor types.

DETAILED DESCRIPTION:
This is an open-label trial of ImmuniCell® treatment of patients with malignant melanoma, renal cell cancer (RCC) or non-small cell lung cancer (NSCLC) which are refractory to current treatment or who have indolent disease for which immunotherapy may be beneficial. The trial is designed to identify a safe dose of ImmuniCell® for future clinical trials, to identify a response signal from one or more of the cancers under investigation and to confirm the safety and efficacy in the selected target tumour.

The trial has three stages:

Stage I comprising a safety cohort of patients to identify a safe dose Stage II comprising an expanded patient group for response signal identification Stage III to confirm efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥18 years
2. Performance status Eastern Cooperative Oncology Group (ECOG) 0 or 1
3. Subjects with histological or cytological confirmation of advanced malignant melanoma, renal cell carcinoma or NSCLC which are refractory to current standard treatments or who have indolent disease for which immunotherapy may be beneficial
4. Measurable disease according to the irRC criteria
5. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted <2 weeks prior to Cycle 1:

   * Creatinine ≤ 1.5 x upper limit of normal (ULN) OR a calculated creatinine clearance ≥ 50 ml/min
   * Total bilirubin ≤ 1.5 x ULN
   * Alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 2.5 x ULN or ≤ 5 x ULN with liver metastases
   * Absolute lymphocyte count ≥1.0 x 10E9/L
   * Absolute Neutrophil Count (ANC) ≥1.5 x 10E9/L
   * Platelets ≥100 x 10E9/L
   * Haemoglobin ≥ 10 g/dL
6. Life expectancy of at least 3 months
7. Suitable increase in starting γδ T cell number to final γδ T cell number in the proliferation assay between 10 days in culture
8. Able to give informed, written consent
9. For female patients and female partners of male patients: must be surgically sterile, postmenopausal, or compliant with two forms of contraception (one of which must be a barrier method) during and for 6 months after the treatment period; female patients must have a negative urine pregnancy test at screening and must not be breast-feeding.

Exclusion Criteria:

1. Other primary cancers apart from non-melanoma skin cancers, carcinoma - in situ of the cervix, or a prior cancer treated with curative intent more than 2 years ago without any evidence or recurrent disease
2. Uncontrolled systemic infection
3. Systemic steroid therapy or other immune-suppressants (except in cases where the patient is receiving treatment with replacement doses for adrenal insufficiency)
4. Treatment with bisphosphonates, for instance zoledronate, in the previous 3 months and throughout the trial
5. New York Heart Association (NYHA) functional class ≥3 or myocardial infarction within 6 months
6. Clinically-significant uncontrolled cardiac arrhythmia other than asymptomatic atrial fibrillation not requiring therapy.
7. Ulcerative Colitis / Inflammatory bowel disease, Addison's disease
8. Pregnancy or lactation before or during the trial. A urine pregnancy test will be carried out at screening
9. Taking any other investigational medicinal product (IMP) or participation in another interventional clinical trial in the previous 30 days
10. Less than 4 weeks since systemic anti-cancer therapy (tyrosine kinase inhibitors, chemotherapy, immunotherapy, hormonal therapy, radiotherapy) and less than 6 weeks since mitomycin C and nitrosureas
11. Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the trial or evaluation of the trial results
12. Any other condition considered by a trial physician to be inappropriate for inclusion to the study such as contraindications to leukapheresis (contraindications to heparin which are: recent cerebral haemorrhage; peptic ulcer; recent surgery to eye or nervous system; hypersensitivity to heparin; past history of Type II heparin induced thrombocytopenia; past history of significant spontaneous haemorrhage; known haemophilia or other bleeding disorder).
13. Serological evidence of active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-12; Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-27 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with drug-related > grade 3 toxicity (except for nausea, vomiting or grade 3 diarrhoea without maximal supportive therapy; anaemia, alopecia, or asymptomatic grade 3 laboratory findings that last for < 7 days) | 3 months
Document the clinical response (immediate or delayed CR, PR, SD or PD) of the patients following ImmuniCell® treatment and assess the data for a response signal to guide the confirmatory stage | 12 months

SECONDARY OUTCOMES:
Changes in markers of immune response (such as IFN-γ, IL-2 and TNF-α) before the first and subsequent ImmuniCell® infusions | 12 months
  Changes in markers of immune response (such as IFN-γ, IL-2 and TNF-α) before the first and subsequent ImmuniCell® infusions
Changes in peripheral T lymphocyte counts before the first and subsequent ImmuniCell® infusions (optional) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Evans, Prof., Principal Investigator — Beatson West of Scotland Cancer Centre, 1053 Great Western Road, Glasgow G12 0YN
Locations (7):
- United Kingdom (7):
  - Velindre Cancer Centre and University Hospital of Wales, Cardiff
  - Western General Hospital, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St. James's University Hospital, Leeds
  - University College London Hospital, London
  - Churchill Hospital, Oxford
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes